CLINICAL TRIAL: NCT03981198
Title: Proof of Concept (POC) Study of the Soliton Rapid Acoustic (RAP) Nov Heavy Device for the Treatment of Cellulite
Brief Title: Proof of Concept (POC) Study of the Soliton Rapid Acoustic (RAP) for the Treatment of Cellulite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soliton (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Soliton 2018-001
Record Dates: First submitted 2019-05-31; First posted 2019-06-10 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Cellulite
MeSH Terms: conditions — Cellulite

STUDY DESIGN:
Intervention Model Description: Single Group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- RAP treatment (Other): Single RAP treatment applied to thigh and multi-treatment applied to the other thigh.
  Interventions: Device: Soliton Rapid Acoustic Pulse (RAP)

INTERVENTIONS:
Device: Soliton Rapid Acoustic Pulse (RAP) — Treatment of legs and/or buttocks for the temporary improvement in the appearance of cellulite.
  Other Names: RAP

SUMMARY:
Feasibility study is to evaluate the safety, tolerability and efficacy of Soliton's Rapid Acoustic Pulse (RAP) device for the treatment of cellulite

DETAILED DESCRIPTION:
To assess the safety and tolerability of Soliton's RAP Nov Heavy for the treatment of cellulite. To assess the efficacy of Soliton's RAP Nov Heavy device for the temporary improvement in appearance of cellulite in terms of mean change in cellulite severity score (CSS).

ELIGIBILITY:
Inclusion Criteria:

* Female ages 18-65 years
* Participant seeking treatment of cellulite in the upper lateral thigh areas
* Participant presenting with cellulite Grade I or II on both thighs as graded using the Nurnberger-Muller scale classification (Appendix A)
* Participant has stable weight. Body Mass Index (B.M.I.) is ≤ 30
* Participant will not have any other cellulite treatments for 12 months before and throughout the 3-month follow-up
* Participant is willing to participate in study and adhere to follow-up schedule
* Participant is able to read and comprehend English
* Participant has completed Informed Consent Form

Exclusion Criteria:

* Participant is pregnant or planning to become pregnant during the duration of the study
* Participant has a BMI > 30
* Greater than 10% increase or decrease in body weight within past 6 months
* Cellulite treatment on the thighs or buttocks in the last 12 months (Topical or non-invasive procedure)
* Metal or plastic implants in the area of the treatment (vascular stent, or implants in the hips, knees, etc.)
* Active electronic implants such as pacemakers, defibrillators, cochlear implants, nerve/brain stimulators, drug pump, etc.
* Prior liposuction in the thighs or buttocks or any other invasive procedure to limit cellulite.
* Medical disorder that would hinder the wound healing or immune response (no blood disorder, diabetes, inflammatory disease, etc.)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 10 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
Incidence of SAEs | 18 weeks
  The primary safety endpoint will be met if all treated Participants are free from serious adverse events (SAEs) attributable to the RAP device immediately post treatment and at the 3-month follow-up visit.
Treatment Tolerability | 18 Weeks
  The primary endpoint will be met if a mean tolerability measure using pain scores averaged across all treated Participants is < 8.0

SECONDARY OUTCOMES:
Cellulite improvement | 18 weeks
  A ≥15% mean reduction in the 0-5-point Cellulite Severity Scale as determined by physician assessment of Participant photographs taken before and 3 months after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher C Capelli, MD, Study Director — Soliton
Locations (1):
- SkinCare Physicians, Chestnut Hill, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No